CLINICAL TRIAL: NCT02983474
Title: Development of Cholecystectomy Complication Predictive Model for Developing the Surgical Quality Improvement Program
Brief Title: Korea Surgical Quality Improvement Program
Acronym: KSQIP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: NH16-007
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cholecystectomy — Laparoscopic surgery
  1. Reverse Trendelenburg position
  2. Skin incision and trocar insertion
  3. CO2 gas insufflation
  4. Intra-abdominal inspection and gallbladder exposure
  5. Gallbladder traction
  6. Calot triangle exposure
  7. Cystic artery and cystic duct isolation
  8. Gallbladder bed dissection
  9. Bleeding control
  10. Gallbladder extraction
  11. Trocar removal and wound closure
  Open surgery
  1. Supine position
  2. Skin incision
  3. Intra-abdominal inspection and gallbladder exposure
  5. Gallbladder traction 6. Calot triangle exposure 7. Cystic artery and cystic duct isolation 8. Gallbladder bed dissection 9. Gallbladder extraction 10. Bleeding control 11. Wound closure

SUMMARY:
The member of National Evidence-based Healthcare Collaborating Agency and the planning committee of Korean Association of hepato-biliary pancreatic Surgery established the protocol of Korean Surgical Quality Improvement Program (KSQIP) with verifying variables of American College of Surgeons - National Surgical Quality Improvement Program (ACS-NSQIP and National Clinical Database (NCD) of Japan; demographics, preoperative information, laboratory values, operation finding, general occurrences, postoperative occurrences, and follow-up data to develop post cholecystectomy complication risk model.

The 50 surgeons from 20 hospitals have decided to participated in the primary prospective study to apply KSQIP to cholecystectomy. The investigators developed web-based database system (http://www.ksqip.org/gb) and surgical clinical reviewer of each hospital will fill out the case report form. Finally, the investigators will provide a risk-adjusted surgical risk calculator and feedback system for reducing complication.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent cholecystectomy with cholecystitis or gallbladder polyp or cholelithiasis

Exclusion Criteria:

* Under 18 age
* Who underwent other abdominal surgery simultaneously
* Gallbladder Cancer, cholangiocarcinoma
* Who did not agree with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who underwent cholecystectomy with cholecystitis or gallbladder polyp or cholelithiasis
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Composite of bile leakage and iatrogenic duct injury | 1 month

IPD SHARING:
Plan to Share IPD: No